CLINICAL TRIAL: NCT03448068
Title: Low-dose Ketamine Infusions for Perioperative Pain Management in Patients Undergoing Laparoscopic Gastric Bypass
Brief Title: Perioperative Ketamine for Pain With Gastric Bypass
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Andrew Gorlin, MD, Assistant Professor of Anesthesiology, College of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-000301
Record Dates: First submitted 2018-02-09; First posted 2018-02-27 (Actual); Results first posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Laparoscopic Gastric Bypass Surgery; Ketamine
MeSH Terms: interventions — Ketamine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine Therapy (Experimental): 1. Ketamine 0.3 mg/kg (IBW) bolus with induction.
  2. Ketamine infusion 0.2 mg/kg/hr. (IBW) initiated after induction and terminated after 24 hours.
  3. Ketamine infusion will not be titrated.
  4. Remaining care will be identical to standard therapy group.
  Interventions: Drug: Ketamine
- Standard Therapy (Active Comparator): 1. Calculation ideal body weight (IBW)
  2. Pre-op dexamethasone
  3. Pre-op midazolam at discretion of anesthesiologist
  4. Anesthesia Induction - Propofol and fentanyl, anesthesiologist discretion. Neuromuscular block with succinylcholine and/or rocuronium at discretion of anesthesiologist. Orotracheal intubation.
  5. Anesthesia Maintenance - Sevoflurane/rocuronium. Addl. doses of fentanyl, discretion of anesthesiologist.
  6. Emergence from anesthesia - Acetaminophen, Ketorolac and Ondansetron unless contraindicated. Sugammadex depending on twitch response per drug manufacturer recommended protocol.
  7. Post-Op Analgesia - Hydromorphone, acetaminophen and ketorolac
  8. Other post-op care as per usual surgical routine
  Interventions: Drug: Standard therapy

INTERVENTIONS:
Drug: Ketamine — Ketamine 0.3 mg/kg (IBW) bolus with induction. Ketamine infusion 0.2mg/kg/hr. (IBW) initiated after induction and terminated after 24 hours.
  Ketamine infusion not titrated.
  Arms: Ketamine Therapy
Drug: Standard therapy — Pre-op dexamethasone 4mg IV and midazolam 1-2mg IV Anesthesia Induction - Propofol 2-3mg/kg IV, Fentanyl 1mcg/kg IV, neuromuscular block w/succinylcholine and/or rocuronium, orotracheal intubation Anesthesia maintenance - Sevoflurane/rocuronium, fentanyl 0.5-1mcg/kg Anesthesia emergence - Acetaminophen 1g, ketorolac 30 mg IV, ondansetron 4mg IV, sugammadex 2mg/kg or 4 mg/kg dose depending on twitch Post-op anesthesia - Hydromorphone patient-controlled analgesia (PCA) 0.2 mg/8 min, acetaminophen 1 g IV Q8 around the clock (ATC) x 3 addl. doses, ketorolac 15 mg IV Q6 ATC x 3 addl. doses.
  Other standard surgical post-op care
  Arms: Standard Therapy

SUMMARY:
Opioid medications such as morphine, hydrocodone and oxycodone are standard for treating pain after surgery, however there are disadvantages. Because of the way opioids work, gastric bypass patients may have an increased risk of having sedation or problems with breathing. In patients with sleep apnea, opioids may increase the risk of severe apnea.

Ketamine is an alternative pain medicine that can be used to treat pain after surgery and may have fewer effects on breathing. Using ketamine as part of the regimen may be a better choice for laparoscopic gastric bypass patients.

This study is being done to find out if intraoperative ketamine infusion combined with continuation for twenty-four hours post-surgery provides superior pain control and decreases post-operative opioid use versus standard non-ketamine therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing laparoscopic gastric bypass at Mayo Clinic in Arizona
2. BMI is ≥ 35 kg/m2
3. Consent is able to be obtained as per Mayo Clinic policy

Exclusion Criteria:

1. Intolerance to ketamine
2. History of schizophrenia, schizoaffective disorder, or other psychiatric diagnosis with psychotic features
3. Presence of unstable cardiovascular disease (presence of acute coronary syndrome, unstable angina, hypertension emergency, acute transient ischemic attack (TIA) or stroke)
4. Presence of acute elevation of intracranial or intraocular pressure
5. Presence of seizure disorder
6. History of substance abuse or addiction
7. Creatinine greater than 1.5 mg/dL
8. End-stage liver disease
9. Pregnancy
10. Patients with chronic pain and/or chronic opioid therapy will not be excluded to more closely replicate the study patient population of interest. However, patients taking greater than 50 morphine equivalents (ME) per day for greater than 1 month prior to surgery will be excluded.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Gorlin, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Phoenix, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketamine Therapy: Subjects received a ketamine bolus (0.3 mg/kg IV IBW) with induction; a ketamine infusion (0.2 mg/kg/hr IBW) was started after induction and terminated the next morning after surgical team rounds or at 24 hours
- Standard Therapy: Subjects received standard of care anesthesia
Period: Overall Study
Arm/Group | Ketamine Therapy | Standard Therapy
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine Therapy | Standard Therapy | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (11.5) | 48.8 (10.2) | 51.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 5 | 2 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Total Cumulative Perioperative Opioid Dose
Description: Measured in oral morphine equivalents
Time Frame: approximately 48 hours after induction of anesthesia
Measure: Mean (Standard Deviation); unit: Morphine Equivalents
Arm/Group | Ketamine Therapy | Standard Therapy
Number analyzed (Participants) | 17 | 17
Morphine Equivalents | 179.9 (113.1) | 248.6 (91.6)
Statistical Analysis 1: Comparison: Ketamine Therapy vs Standard Therapy; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Average Pain Score 0-12 Hours
Description: Patient reported pain scores at 0-12 hours post operatively. Measured by a 100 mm long Visual Analog Scale (VAS). The VAS does not have any pre-set marks between the extremes of 0 for no pain and 100 mm for extreme pain. The investigator measures the mark made by the participant in mm and records this for the value of pain. A higher score indicates great pain intensity.
Time Frame: approximately 0-12 hours post operatively
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ketamine Therapy | Standard Therapy
Number analyzed (Participants) | 17 | 17
mm | 3.4 (2.2) | 4.2 (1.5)
Statistical Analysis 1: Comparison: Ketamine Therapy vs Standard Therapy; Test type: Superiority; p = 0.2252, t-test, 2 sided

3. Secondary Outcome: Average Pain Score 12-24 Hours
Description: Patient reported pain scores at 12-24 hours post operatively. Measured by a 100 mm long Visual Analog Scale (VAS). The VAS does not have any pre-set marks between the extremes of 0 for no pain and 100 mm for extreme pain. The investigator measures the mark made by the participant in mm and records this for the value of pain. A higher score indicates great pain intensity.
Time Frame: approximately 12-24 hours post operatively
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ketamine Therapy | Standard Therapy
Number analyzed (Participants) | 17 | 17
mm | 2.6 (1.9) | 3.7 (1.4)
Statistical Analysis 1: Comparison: Ketamine Therapy vs Standard Therapy; Test type: Superiority; p = 0.0610, t-test, 2 sided

4. Secondary Outcome: Average Pain Score 24-48 Hours
Description: Patient reported pain scores at 24-48 hours post operatively. Measured by a 100 mm long Visual Analog Scale (VAS). The VAS does not have any pre-set marks between the extremes of 0 for no pain and 100 mm for extreme pain. The investigator measures the mark made by the participant in mm and records this for the value of pain. A higher score indicates great pain intensity.
Time Frame: approximately 24-48 hours post operatively
Population: 2 subjects were discharged early so data was not collected or analyzed for 1 subject from the ketamine therapy group and 1 subject from the standard therapy group
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ketamine Therapy | Standard Therapy
Number analyzed (Participants) | 16 | 16
mm | 3.1 (1.9) | 3.8 (1.5)
Statistical Analysis 1: Comparison: Ketamine Therapy vs Standard Therapy; Test type: Superiority; p = 0.2720, t-test, 2 sided

5. Secondary Outcome: Post-Operative Nausea
Description: Number of subject to experience post-operative nausea
Time Frame: 12 hours, 24 hours, and 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Therapy | Standard Therapy
Number analyzed (Participants) | 17 | 17
Participants
  Nausea 1st 12 hours | 10 | 9
  Nausea 2nd 12 hours | 6 | 2
  Nausea 2nd 24 hours | 3 | 3
Statistical Analysis 1: Comparison: Ketamine Therapy vs Standard Therapy; Nausea 1st 12 hours for Ketamine Therapy vs Standard Therapy; Test type: Superiority; p = 0.7298, Chi-squared
Statistical Analysis 2: Comparison: Ketamine Therapy vs Standard Therapy; Nausea 2nd 12 hours for Ketamine Therapy vs Standard Therapy; Test type: Superiority; p = 0.1058, Chi-squared
Statistical Analysis 3: Comparison: Ketamine Therapy vs Standard Therapy; Nausea 2nd 24 hours for Ketamine Therapy vs Standard Therapy; Test type: Superiority; p = 1.000, Chi-squared

6. Secondary Outcome: Length of Stay in Hospital
Description: Length of hospital stay measured in hours
Time Frame: Arrival at hospital until discharge from hospital, approximately 2 days
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Ketamine Therapy | Standard Therapy
Number analyzed (Participants) | 17 | 17
Hours | 43.9 (18.0) | 36.7 (14.0)
Statistical Analysis 1: Comparison: Ketamine Therapy vs Standard Therapy; Test type: Superiority; p = 0.2, t-test, 2 sided

7. Secondary Outcome: Patient Satisfaction With Pain Control at Time of Hospital Discharge
Description: Self-reported questionnaire at the time of discharge from the hospital rating satisfaction of pain treatment while in the hospital using a scale of 0= extremely dissatisfied, 10 = extremely satisfied.
Time Frame: approximately 1-2 days post-operatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine Therapy | Standard Therapy
Number analyzed (Participants) | 17 | 17
score on a scale | 9.5 (0.9) | 8.3 (1.9)

8. Secondary Outcome: Patient Satisfaction With Pain Control at Postoperative Visit
Description: Self-reported questionnaire at the time of first post-operative visit with the surgeon, rating the worst amount of pain since being discharged from the hospital using a scale of 0= no pain, 10 = worst pain possible.
Time Frame: approximately 30 days post-operatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketamine Therapy | Standard Therapy
Number analyzed (Participants) | 17 | 17
score on a scale | 3.6 (3.4) | 6.2 (2.3)

ADVERSE EVENTS:
Time Frame: Adverse events were collected 30 days following surgery for each participant, over a study duration of approximately 48 months
Arm/Group | Ketamine Therapy | Standard Therapy
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 13/17 | 11/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine Therapy (N=17) | Standard Therapy (N=17)
Nausea (General disorders) | 13 (19) | 11 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT03448068/Prot_SAP_000.pdf